CLINICAL TRIAL: NCT01898884
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Multicenter, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Oral VP 20629 in Adult Subjects With Friedreich's Ataxia
Brief Title: Safety and Pharmacology Study of VP 20629 in Adults With Friedreich's Ataxia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20629-100
Record Dates: First submitted 2013-07-03; First posted 2013-07-15 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Friedreich's Ataxia
MeSH Terms: conditions — Friedreich Ataxia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose of VP 20629 or placebo (Experimental): Four groups of 8 subjects each will receive a single dose of VP 20629 (150 mg, 450 mg, 900 mg, or 1200 mg) or placebo.
  Interventions: Drug: VP 20629; Drug: Placebo
- Multiple doses of VP 20629 or placebo (Experimental): Three groups of 8 subjects each will receive multiple doses of VP 20629 (300 mg, 600 mg, or 900 mg total daily dose) or placebo. VP 20629 or placebo will be administered every 8 hours for 7 days with a single morning dose on Day 8.
  Interventions: Drug: VP 20629; Drug: Placebo

INTERVENTIONS:
Drug: VP 20629
  Other Names: Indole-3-propionic acid
Drug: Placebo

SUMMARY:
The objectives of the study are:

* To evaluate the safety and tolerability of single and multiple oral doses of VP 20629 in subjects with Friedreich's ataxia (FA). [Primary]
* To characterize the pharmacokinetics of VP 20629 by investigation of the plasma concentration-time profile following single and multiple oral doses in subjects with FA. [Secondary]
* To investigate the pharmacodynamic effects of VP 20629 on plasma 8-isoprostane and malondialdehyde and urinary 8-hydroxydeoxyguanosine concentrations following multiple oral doses in subjects with FA. [Exploratory]

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 to 45 years of age (inclusive).
2. Have a body mass index between 18 and 27 kg/m^2 (inclusive).
3. Have a clinical presentation consistent with FA.
4. Have a confirmed diagnosis of FA with a defined expanded guanosine, adenine, adenine (GAA) triplet repeat number.
5. Have an International Cooperative Ataxia Rating Scale (ICARS) mean total score of ≤75.
6. If female, be postmenopausal (cessation of menses ≥1 year), surgically sterile, or have a negative serum human chorionic gonadotropin pregnancy test within 5 days prior to the first dose of study drug. Women of child bearing potential must also be on an acceptable method of birth control, as determined by the Investigator, for 3 months prior to the first dose and must agree to continue use through 2 months after the last dose of study drug.

   If male, be surgically sterile or agree to follow an acceptable method of birth control as determined by the Investigator, from the screening visit through 2 months after the last dose of study drug.
7. Be able to swallow capsules whole.
8. Agree to adhere to the protocol-defined schedule of assessments and procedures.
9. Be informed of the nature of the study and provide written informed consent before any study-specific procedures are performed.

Exclusion Criteria:

1. Have taken coenzyme Q10, idebenone, other dietary or herbal supplements (with an anti-oxidative effect), or over-the-counter medications (including homeopathic medicines and vitamins) within 1 week prior to the first dose of study drug on Day 1.
2. If female, be pregnant or breastfeeding.
3. Have a positive test result for human immunodeficiency virus (HIV), hepatitis B surface antigen, or hepatitis C antibody.
4. Have ingested any alcohol within 48 hours before admission to the clinical study unit on Day -1. NOTE: Caffeine intake should be limited to 2 caffeine-containing beverages per day during this same time period.
5. Have participated in an investigational drug trial within 30 days prior to the first dose of study drug on Day 1. NOTE: Subjects who received study drug (VP 20629 or placebo) in a single-dose group in this study and completed the Post-treatment Safety Assessment are allowed to enroll in a multiple-dose group following a 21 day washout period, provided they continue to meet protocol eligibility criteria. Subjects cannot enroll in a multiple-dose group if they have an ongoing adverse event following participation in a single-dose group or had a serious adverse event during a single-dose group (regardless of causality).
6. Have a known hypersensitivity to any ingredient in the study formulation.
7. Have, as determined by the Investigator and/or medical monitor, any clinically relevant medical or surgical condition that could interfere with the administration of study drug, interpretation of study results, or compromise the safety or well-being of the subject.
8. Have a Columbia-Suicide Severity Rating Scale (C-SSRS) score of 4 or 5.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2013-08-13 (Actual); Primary Completion 2015-06-18 (Actual); Study Completion 2015-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- United States (5):
  - UCLA Medical Center, Los Angeles, California
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multicenter study conducted between 13 August 2013 and 18 June 2015.
Pre-assignment Details: A total of 46 participants were enrolled to the study, of which 32 were randomly assigned to single-dose group and 24 were randomly assigned to multiple-dose group. Participants who received investigational product in a single-dose group and completed the post-treatment safety assessment were allowed to enrol in a multiple-dose group.
Groups:
- Single Dose Placebo: Participants received placebo matching to single dose of VP 20629 capsules orally under fasting condition on Day 1.
- Single Dose VP 20629 150 mg: Participants received single dose of VP 20629 capsules of 150 milligram (mg) orally under fasting condition on Day 1.
- Single Dose VP 20629 450 mg: Participants received single dose of VP 20629 capsules of 450 mg orally under fasting condition on Day 1.
- Single Dose VP 20629 900 mg: Participants received single dose of VP 20629 capsules of 900 mg orally under fasting condition on Day 1.
- Single Dose VP 20629 1200 mg: Participants received single dose of VP 20629 capsules of 1200 mg orally under fasting condition on Day 1.
- Multiple Dose Placebo: Participants received placebo matching to multiple doses of VP 20629 capsules orally daily from Day 1 to Day 8 morning under fasting conditions.
- Multiple Dose VP 20629 300 mg: Participants received VP 20629 capsules 300 mg total daily dose in 3 divided doses (100 mg every 8 hours) orally daily from Day 1 to Day 8 morning under fasting conditions.
- Multiple Dose VP 20629 600 mg: Participants received VP 20629 capsules 600 mg total daily dose in 3 divided doses (200 mg every 8 hours) orally daily from Day 1 to Day 8 morning under fasting conditions.
- Multiple Dose VP 20629 900 mg: Participants received VP 20629 capsules 900 mg total daily dose in 3 divided doses (300 mg every 8 hours) orally daily from Day 1 to Day 8 morning under fasting conditions.
Period: Single Dose Period
Arm/Group | Single Dose Placebo | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg | Multiple Dose Placebo | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Started | 8 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0
Completed | 8 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Multiple Dose Period
Arm/Group | Single Dose Placebo | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg | Multiple Dose Placebo | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Started | 0 | 0 | 0 | 0 | 0 | 6 (Eligible participants who completed single dose treatment were randomized to multiple dose groups.) | 6 (Eligible participants who completed single dose treatment were randomized to multiple dose groups.) | 6 (Eligible participants who completed single dose treatment were randomized to multiple dose groups.) | 6 (Eligible participants who completed single dose treatment were randomized to multiple dose groups.)
Treated | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Randomized Not Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) set consisted of all participants who were randomly assigned to an investigational product treatment group. The baseline data for 14 participants who were randomised directly to multiple dose groups, was not summarised and not reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Dose Placebo | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.1 (7.04) | 22.7 (1.97) | 27.8 (4.45) | 28.0 (6.90) | 26.8 (8.86) | 26.0 (6.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 2 | 3 | 4 | 17
  Male | 3 | 3 | 4 | 3 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs (TEAEs), defined as all AEs that start during study drug treatment (and up to 7 days after the last dose of the study drug) and were not seen at baseline, or were seen at baseline but increased in frequency and/or severity during study drug treatment (and up to 7 days after the last dose of study drug).
Time Frame: From Start of Study Treatment up to Day 19
Population: The ITT-safety (ITT-S) set consisted of all participants who were randomly assigned to an investigational product treatment group and who received at least 1 partial or complete dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Single Dose Placebo | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg | Multiple Dose Placebo | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5
participants
  TEAE | 3 | 0 | 4 | 5 | 6 | 4 | 3 | 6 | 3
  TESAE | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities Recorded as Treatment-Emergent Adverse Events (TEAEs)
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation were reported as an adverse event. Treatment-emergent were events between first dose of study drug and 7 days after the last dose that were absent before treatment or that worsened relative to pretreatment state. Number of participants with Grade 3 or higher treatment-emergent adverse events for laboratory abnormalities were reported as clinically relevant laboratory changes.
Time Frame: From Start of Study Treatment up to Day 19
Population: The ITT-S set consisted of all participants who were randomly assigned to an investigational product treatment group and who received at least 1 partial or complete dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Single Dose Placebo | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg | Multiple Dose Placebo | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5
participants
  Blood Glucose Increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants With Vital Signs Abnormalities Recorded as Treatment-Emergent Adverse Events (TEAEs)
Description: Vital sign assessments included systolic blood pressure, diastolic blood pressure, heart rate, and temperature. Vital signs abnormalities reported as TEAEs were reported.
Time Frame: From Start of Study Treatment up to Day 19
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- Single Dose VP 20629 450 mg: Participants received single dose VP 20629 capsules of 450 mg orally under fasting condition on Day 1.
- Single Dose VP 20629 900 mg: Participants received single dose VP 20629 capsules of 900 mg orally under fasting condition on Day 1.
- Single Dose VP 20629 1200 mg: Participants received single dose VP 20629 capsules of 1200 mg orally under fasting condition on Day 1.
Arm/Group | Single Dose Placebo | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg | Multiple Dose Placebo | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Relevant Electrocardiogram (ECG) Abnormalities Recorded as Adverse Events (AEs)
Description: ECG included PR interval, QRS interval, QTcB interval, QTcF interval were considered as clinically significant ECG abnormalities.
Time Frame: From Start of Study Treatment up to Day 19
Population: as for outcome 2
Measure: Number; unit: participants
Groups:
- Single Dose VP 20629 150 mg: Participants received single dose VP 20629 capsules of 150 milligram (mg) orally under fasting condition on Day 1.
Arm/Group | Single Dose Placebo | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg | Multiple Dose Placebo | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5
participants | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

5. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of VP 20629 and Its Metabolite (VP 20631) for Single Dose Groups
Description: The Cmax is the maximum observed plasma concentration of single dose of VP 20629 and VP 20631.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8,10, 12, 24 and 48 hours Postdose on Day 1
Population: The pharmacokinetic set consisted of participants who had quantifiable VP 20629 plasma concentrations. Here, "N" (Number of participants analyzed) and "n" are number of participants analyzed for this outcome measure and for the specified compound, respectively.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Single Dose Placebo | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL)
  VP 20629 (n=7,6,6,6,6) | 269 (92) | 29350 (6344) | 47350 (12742) | 76983 (7293) | 73717 (14848)
  VP 20631 (n=6,6,6,6,6) | 7 (2) | 1068 (353) | 3556 (2347) | 12515 (6056) | 15842 (12438)

6. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of VP 20629 and Its Metabolite (VP 20631) for Single Dose Groups
Description: The Tmax is the time to reach maximum observed plasma concentration of single dose of VP 20629 and VP 20631.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8,10, 12, 24 and 48 hours Postdose on Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Single Dose Placebo | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 6
hour
  VP 20629 (n=7,6,6,6,6) | 9.94 (7.58) | 1.50 (0.45) | 1.92 (0.95) | 1.83 (0.61) | 3.01 (1.77)
  VP 20631(n=6,6,6,6,6) | 23.71 (20.17) | 2.17 (0.41) | 2.83 (2.50) | 2.16 (0.60) | 3.35 (2.33)

7. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of VP 20629 and Its Metabolite (VP 20631) for Single Dose Groups
Description: The AUC is the area under the plasma concentration-time curve observed.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8,10, 12, 24 and 48 hours Postdose on Day 1
Population: The pharmacokinetic set consisted of participants who had quantifiable VP 20629 plasma concentrations.
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour*nanogram per milliliter (h*ng/mL)
  VP 20629 | 152277 (27113) | 298443 (42925) | 463893 (44896) | 525976 (107856)
  VP 20631 | 5118 (1155) | 14208 (4117) | 33366 (9374) | 48322 (17989)

8. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC[0-8]) of VP 20629 and Its Metabolite (VP 20631) for Single Dose Groups
Description: The AUC(0-8) is the area under the plasma concentration-time curve from time zero to 8 hours postdose.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, and 8 hours Postdose on Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Single Dose VP 20629 150mg: Participants received single dose VP 20629 capsules of 150 milligram (mg) orally under fasting condition on Day 1.
Arm/Group | Single Dose Placebo | Single Dose VP 20629 150mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 6
h*ng/mL
  VP 20629 (n=7,6,6,6,6) | 1708 (693) | 95673 (10720) | 183398 (10155) | 302823 (31529) | 325019 (45937)
  VP 20631 (n=5,6,6,6,6) | 21 (27) | 3201 (802) | 9934 (4155) | 27426 (8969) | 37258 (19280)

9. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve to the Last Measurable Plasma Concentration (AUCt) of VP 20629 and Its Metabolite (VP 20631) for Single Dose Groups
Description: The AUCt is the measure of the plasma drug concentration from time zero to time t.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8,10, 12, 24 and 48 hours Postdose on Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Single Dose Placebo | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 6
h*ng/mL
  VP 20629 (n=7,6,6,6,6) | 9903 (4192) | 147287 (25078) | 294510 (41445) | 457563 (46848) | 519996 (106355)
  VP 20631 (n=6,6,6,6,6) | 164 (149) | 4876 (1201) | 14070 (4110) | 33121 (9322) | 48114 (17934)

10. Secondary Outcome: Terminal Plasma Half-Life (t1/2) of VP 20629 and Its Metabolite (VP 20631) for Single Dose Groups
Description: The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8,10, 12, 24 and 48 hours Postdose on Day 1
Population: The pharmacokinetic set consisted of participants who had quantifiable VP 20629 plasma concentrations.
Measure: Median (Full Range); unit: hour
Arm/Group | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour
  VP 20629 | 9.98 [8.46 to 13.56] | 7.87 [7.62 to 8.46] | 7.43 [4.40 to 9.44] | 7.85 [6.62 to 8.97]
  VP 20631 | 11.19 [9.14 to 15.09] | 7.85 [7.13 to 8.22] | 7.72 [4.52 to 9.46] | 6.95 [6.29 to 8.52]

11. Secondary Outcome: Volume of Distribution (Vz/F) of VP 20629 for Single Dose Groups
Description: The Vz is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8,10, 12, 24 and 48 hours Postdose on Day 1
Population: The pharmacokinetic set consisted of participants who had quantifiable VP 20629 plasma concentrations.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Liter | 15.0 (3.4) | 17.6 (2.9) | 20.8 (6.1) | 26.9 (6.3)

12. Secondary Outcome: Total Body Drug Clearance (CL/F) of VP 20629 for Single Dose Groups
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8,10, 12, 24 and 48 hours Postdose on Day 1
Population: The pharmacokinetic set consisted of participants who had quantifiable VP 20629 plasma concentrations.
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
liter per hour | 1.010 (0.171) | 1.533 (0.209) | 1.956 (0.196) | 2.357 (0.447)

13. Secondary Outcome: Elimination Rate Constant (Lambda[z]) of VP 20629 and Its Metabolite (VP 20631) for Single Dose Groups
Description: Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8,10, 12, 24 and 48 hours Postdose on Day 1
Population: The pharmacokinetic set consisted of participants who had quantifiable VP 20629 plasma concentrations.
Measure: Mean (Standard Deviation); unit: per hour
Arm/Group | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
per hour
  VP 20629 | 0.0688 (0.0111) | 0.0874 (0.0033) | 0.1007 (0.0312) | 0.0892 (0.0105)
  VP 20631 | 0.0615 (0.0114) | 0.0889 (0.0046) | 0.0958 (0.0295) | 0.0972 (0.0124)

14. Secondary Outcome: Cumulative Amount Excreted Into the Urine (Ae) for Unchanged VP 20629 and Its Metabolite (VP 20631) for Single Dose Groups
Description: The Ae is the amount of drug excreted in urine. It is calculated by multiplying the urinary volume with the urinary drug concentration.
Time Frame: 0-4, 4-8, 8-16, 16-24, 24-36 and 36-48 hours postdose on Day 1
Population: The pharmacokinetic set consisted of participants who had quantifiable VP 20629 plasma concentrations. Here, "N" is number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: microgram (mcg)
Arm/Group | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg
Number analyzed (Participants) | 4 | 4 | 5 | 5
microgram (mcg)
  VP 20629 | 55.0 (17.2) | 79.4 (13.3) | 368.6 (196.3) | 518.1 (105.6)
  VP 20631 | 131644.9 (19834.5) | 529022.1 (92223.8) | 953370.1 (116994.6) | 1263419.7 (190242.9)

15. Secondary Outcome: Percentage of Drug Excreted in Urine (Ae%) of VP 20629 for Single Dose Groups
Description: The Ae% is the percentage of drug dose excreted into the urine calculated as (Ae divided by dose)∗100.
Time Frame: -4, 4-8, 8-16, 16-24, 24-36 and 36-48 hours postdose on Day 1
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg
Number analyzed (Participants) | 4 | 4 | 5 | 5
percentage of dose | 0.0367 (0.0115) | 0.0176 (0.0030) | 0.0410 (0.0218) | 0.0432 (0.0088)

16. Secondary Outcome: Renal Clearance (CLR) of VP 20629 for Single Dose Groups
Description: The CLR is the renal clearance of the drug, calculated as Ae/AUC(0-infinity) on Day 1 or Ae(0-24)/AUC(0-24) on Day 1.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8,10, 12, 24 and 48 hours Postdose on Day 1
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Single Dose VP 20629 150 mg | Single Dose VP 20629 450 mg | Single Dose VP 20629 900 mg | Single Dose VP 20629 1200 mg
Number analyzed (Participants) | 4 | 4 | 5 | 5
liter per hour | 0.0003 (0.0001) | 0.0003 (0.0001) | 0.0008 (0.0005) | 0.0010 (0.0002)

17. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of VP 20629 and Its Metabolite (VP 20631) for Multiple Dose Groups
Description: The Cmax is the maximum observed plasma concentration of Multiple Dose of VP 20629 and VP 20631.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 24 and 72 hours Postdose on Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Multiple Dose Placebo | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5
nanogram per milliliter (ng/mL)
  VP 20629 (n=6,6,6,5) | 172 (82) | 21667 (2890) | 30000 (5592) | 40440 (8878)
  VP 20631 (n=1,6,6,5) | 6 (NA) — Standard deviation was not evaluable as only 1 participant was analyzed. | 556 (88) | 1270 (446) | 2094 (480)

18. Secondary Outcome: Maximum Observed Serum Concentration at Steady State (Cmax,ss) of VP 20629 and Its Metabolite (VP 20631) for Multiple Dose Groups
Description: The Cmax,ss is the maximum observed plasma concentration at steady state.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 and 48 hours Postdose on Day 8
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Multiple Dose Placebo | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5
ng/mL
  VP 20629 (n=6,5,6,5) | 212 (54) | 25060 (10656) | 32583 (6941) | 45000 (3431)
  VP 20631 (n=4,5,6,5) | 5 (3) | 754 (194) | 1638 (252) | 3156 (1305)

19. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of VP 20629 and Its Metabolite (VP 20631) for Multiple Dose Groups
Description: The Tmax is the time to reach maximum observed plasma concentration of multiple dose of VP 20629 and VP 20631.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 24 and 72 hours Postdose on Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Multiple Dose Placebo | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5
hour
  VP 20629 (n=6,6,6,5) | 3.24 (1.72) | 1.09 (0.38) | 1.42 (0.38) | 1.63 (0.71)
  VP 20631 (n=1,6,6,5) | 0.58 (NA) — Standard deviation was not evaluable as only 1 participant was analyzed. | 1.42 (0.49) | 1.59 (0.38) | 2.02 (0.82)

20. Secondary Outcome: Time of Maximum Observed Plasma Concentration at Steady State (Tmax,ss) of VP 20629 and Its Metabolite (VP 20631) for Multiple Dose Groups
Description: The Tmax,ss is the time to reach maximum observed plasma concentration at steady state of multiple dose of VP 20629 and VP 20631.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 and 48 hours Postdose on Day 8
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Multiple Dose Placebo | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 6 | 5 | 6 | 5
hour
  VP 20629 (n=6,5,6,5) | 6.65 (3.96) | 0.97 (0.04) | 2.00 (0.32) | 1.80 (0.91)
  VP 20631 (n=4,5,6,5) | 0.50 (0.71) | 1.67 (0.42) | 2.26 (0.53) | 1.90 (0.89)

21. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of VP 20629 and Its Metabolite (VP 20631) for Multiple Dose Groups
Description: The AUC is the area under the plasma concentration-time curve observed.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 and 48 hours Postdose on Day 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 5 | 6 | 5
h*ng/ml
  VP 20629 | 184407 (108180) | 217115 (58417) | 332140 (73876)
  VP 20631 | 5156 (1869) | 9299 (2402) | 14807 (2206)

22. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve at Steady State (AUCss) of VP 20629 and Its Metabolite (VP 20631) for Multiple Dose Groups
Description: The AUCss is the area under the plasma concentration time curve observed during a dosing at steady state.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, and 8 hours Postdose on Day 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 5 | 6 | 5
h*ng/ml
  VP 20629 | 99794 (44105) | 138567 (37102) | 196587 (18647)
  VP 20631 | 2848 (677) | 6006 (1215) | 9732 (1932)

23. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC[0-8]) of VP 20629 and Its Metabolite (VP 20631) for Multiple Dose Groups
Description: The AUC(0-8) is the area under the plasma concentration-time curve from time zero to 8 hours postdose.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6 and 8 hours Postdose on Day 1
Population: The pharmacokinetic set consisted of participants who had quantifiable VP 20629 plasma concentrations. Here, "n" is number of participants analyzed for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Multiple Dose Placebo | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5
h*ng/mL
  VP 20629 (n=6,6,6,5) | 1080 (451) | 72054 (21395) | 113510 (26091) | 144059 (10302)
  VP 20631 (n=1,6,6,5) | 20 (NA) — Standard deviation was not evaluable as only 1 participant was analyzed. | 1926 (315) | 4130 (1137) | 5740 (1076)

24. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUCt) of VP 20629 and Its Metabolite (VP 20631) for Multiple Dose Groups
Description: The AUCtau is the measure of the plasma drug concentration from time zero to time t.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 and 48 hours Postdose on Day 8
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Multiple Dose Placebo | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 6 | 5 | 6 | 5
h*ng/mL
  VP 20629 (n=6,5,6,5) | 6769 (1480) | 177487 (102429) | 212568 (57087) | 325464 (72038)
  VP 20631 (n=4,5,6,5) | 81 (124) | 4992 (1790) | 9103 (2358) | 14570 (2177)

25. Secondary Outcome: Terminal Plasma Half-Life (t1/2) of VP 20629 and Its Metabolite (VP 20631) for Multiple Dose Groups
Description: as for outcome 10
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 and 48 hours Postdose on Day 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 5 | 6 | 5
hour
  VP 20629 | 9.95 (1.09) | 9.07 (1.21) | 9.05 (1.18)
  VP 20631 | 10.01 (0.44) | 9.68 (1.45) | 9.11 (0.96)

26. Secondary Outcome: Volume of Distribution (Vz/F) of VP 20629 for Multiple Dose Groups
Description: as for outcome 11
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 and 48 hours Postdose on Day 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 5 | 6 | 5
liter | 16.05 (5.28) | 19.77 (4.62) | 20.03 (2.98)

27. Secondary Outcome: Total Body Drug Clearance at Steady State (CLss/F) of VP 20629 for Multiple Dose Groups
Description: as for outcome 12
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 and 48 hours Postdose on Day 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 5 | 6 | 5
liter per hour | 1.133 (0.388) | 1.524 (0.364) | 1.537 (0.140)

28. Secondary Outcome: Elimination Rate Constant (Lambda[z]) of VP 20629 and Its Metabolite (VP 20631) for Multiple Dose Groups
Description: as for outcome 13
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 and 48 hours Postdose on Day 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: per hour
Arm/Group | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 5 | 6 | 5
per hour
  VP 20629 | 0.0703 (0.0076) | 0.0775 (0.0094) | 0.0777 (0.0111)
  VP 20631 | 0.0693 (0.0031) | 0.0729 (0.0107) | 0.0768 (0.0085)

29. Secondary Outcome: Cumulative Amount Excreted Into the Urine at Steady State (Ae,ss) of Unchanged VP 20629 and Its Metabolite (VP 20631) for Multiple Dose Groups
Description: The Ae,ss is the amount of drug excreted in urine. It is calculated by multiplying the urinary volume with the urinary drug concentration.
Time Frame: 0-4, 4-8, 8-16, 16-24, 24-36, and 36-48 hours postdose on Day 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: microgram
Arm/Group | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 5 | 4 | 4
microgram
  VP 20629 | 56.8 (48.1) | 111.4 (27.5) | 244.3 (226.6)
  VP 20631 | 110042 (10852) | 254540 (52440) | 283873 (78764)

30. Secondary Outcome: Percentage of Drug Excreted in Urine at Steady-State (Ae%,ss) of VP 20629 for Multiple Dose Groups
Description: The Ae%,ss is the percentage of drug dose excreted into the urine calculated as (Ae divided by dose)∗100.
Time Frame: 0-4, 4-8, 8-16, 16-24, 24-36, and 36-48 hours postdose on Day 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 5 | 4 | 4
percentage of dose | 0.0568 (0.0481) | 0.0557 (0.0138) | 0.0814 (0.0755)

31. Secondary Outcome: Renal Clearance at Steady State (CLR,ss) of VP 20629 for Multiple Dose Groups
Description: The CLR,ss is the renal clearance of the drug, calculated as Ae/AUC(0-infinity) on Day 8.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24 and 48 hours Postdose on Day 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Multiple Dose VP 20629 300 mg | Multiple Dose VP 20629 600 mg | Multiple Dose VP 20629 900 mg
Number analyzed (Participants) | 5 | 4 | 4
liter per hour | 0.0005 (0.0002) | 0.0009 (0.0004) | 0.0013 (0.0013)

ADVERSE EVENTS:
Time Frame: From the start of the study drug administration upto 30 days after the last dose of study drug administration.
Groups:
- Single Dose Placebo: Participants received placebo matching to single dose of VP 20629 capsules orally under fasting conditions on Day 1.
- Single Dose VP 20629 150mg: Participants received single dose VP 20629 capsules of 150 milligram (mg) orally under fasting conditions on Day 1.
- Single Dose VP 20629 450mg: Participants received single dose VP 20629 capsules of 450 mg orally under fasting conditions on Day 1.
- Single Dose VP 20629 900mg: Participants received single dose VP 20629 capsules of 900 mg orally under fasting conditions on Day 1.
- Single Dose VP 20629 1200mg: Participants received single dose VP 20629 capsules of 1200 mg orally under fasting conditions on Day 1.
- Multiple Dose VP 20629 300mg: Participants received VP 20629 capsules 300 mg total daily dose in 3 divided doses (100 mg every 8 hours) orally daily from Day 1 to Day 8 morning under fasting conditions.
- Multiple Dose VP 20629 600mg: Participants received VP 20629 capsules 600 mg total daily dose in 3 divided doses (200 mg every 8 hours) orally daily from Day 1 to Day 8 morning under fasting conditions.
- Multiple Dose VP 20629 900mg: Participants received VP 20629 capsules 900 mg total daily dose in 3 divided doses (300 mg every 8 hours) orally daily from Day 1 to Day 8 morning under fasting conditions.
Arm/Group | Single Dose Placebo | Single Dose VP 20629 150mg | Single Dose VP 20629 450mg | Single Dose VP 20629 900mg | Single Dose VP 20629 1200mg | Multiple Dose Placebo | Multiple Dose VP 20629 300mg | Multiple Dose VP 20629 600mg | Multiple Dose VP 20629 900mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 1/6 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 3/8 | 0/6 | 4/6 | 5/6 | 6/6 | 4/6 | 3/6 | 6/6 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Dose Placebo (N=8) | Single Dose VP 20629 150mg (N=6) | Single Dose VP 20629 450mg (N=6) | Single Dose VP 20629 900mg (N=6) | Single Dose VP 20629 1200mg (N=6) | Multiple Dose Placebo (N=6) | Multiple Dose VP 20629 300mg (N=6) | Multiple Dose VP 20629 600mg (N=6) | Multiple Dose VP 20629 900mg (N=5)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Dose Placebo (N=8) | Single Dose VP 20629 150mg (N=6) | Single Dose VP 20629 450mg (N=6) | Single Dose VP 20629 900mg (N=6) | Single Dose VP 20629 1200mg (N=6) | Multiple Dose Placebo (N=6) | Multiple Dose VP 20629 300mg (N=6) | Multiple Dose VP 20629 600mg (N=6) | Multiple Dose VP 20629 900mg (N=5)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution may publish results generated from the site individually.